CLINICAL TRIAL: NCT05306899
Title: A Multi-center Randomized Controlled Trial of Efficacy and Safety of Intravenous Ketamine for Chronic Daily Headaches: The KetHead Study
Brief Title: Multi-center RCT of IV Ketamine Efficacy and Safety in Chronic Daily Headaches
Acronym: KetHead
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Canadian Pain Society (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-5523
Record Dates: First submitted 2022-03-02; First posted 2022-04-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10

CONDITIONS: Chronic Daily Headache
Keywords: ketamine; migraine; daily headache; chronic pain
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Chronic Pain | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine infusion (Active Comparator): Intravenous Ketamine
  Interventions: Drug: Ketamine
- Placebo infusion (Placebo Comparator)
  Interventions: Other: 0.9% Saline

INTERVENTIONS:
Drug: Ketamine — Bolus of IV Ketamine 1 mg.kg-1 (= 0.1 ml.kg-1) followed by Infusion of Ketamine 1 mg.kg-1.hour-1 (= 0.5 mL.kg-1.hour-1) for 6 hours. All patients will receive IV midazolam 0.04 mg.kg-1 (maximum 3 mg) and subsequently 0.01-0.02 mg.kg-1 every hour to keep participants in a sedated but arousable state (Ramsay Sedation Scale score 3 or 4) to blind the participants and assessors to group allocation. Ondansetron 8 mg and 8 mg of dexamethasone will be administered to prevent nausea, 5000 units of heparin will be given subcutaneously to prevent thrombo-embolic events.
  Other Names: Ketamine hydrochloride
  Arms: Ketamine infusion
Other: 0.9% Saline — Bolus of IV Saline 0.9% of 0.1 ml.kg-1 followed by Infusion of Saline 0.9% of 0.5 mL.kg-1.hour-1 for 6 hours. All patients will receive IV midazolam 0.04 mg.kg-1 (maximum 3 mg) and subsequently 0.01-0.02 mg.kg-1 every hour to keep participants in a sedated but arousable state (Ramsay Sedation Scale score 3 or 4) to blind the participants and assessors to group allocation. Ondansetron 8 mg and 8 mg of dexamethasone will be administered to prevent nausea, 5000 units of heparin will be given subcutaneously to prevent thrombo-embolic events.
  Other Names: Normal saline
  Arms: Placebo infusion

SUMMARY:
Chronic daily headaches (CDH) poses a significant burden on patients, healthcare systems and the society. Intravenous (IV) ketamine infusion, an intervention that is widely available and scalable, can treat CDH by reversing receptor-mediated sensitization. This study is a multicenter, placebo-controlled, parallel group randomized trial with blinding of participants and observers with the goal of comprehensively assessing the effect of high-dose IV ketamine infusion (1 mg.kg-1.h-1 for six hours) on the frequency and intensity of headaches, mood, activity, sleep, quality of life and safety of ketamine for three months after the interventions. Use of validated questionnaires, wearable technology, a research team that includes investigators with expertise in studying ketamine and in evaluating treatments for CDH and pain syndromes are some of the unique features of this project.

Our study aims to prospectively assess the efficacy and safety of high-dose intravenous ketamine infusions compared to saline infusions in participants with CDH syndrome.

DETAILED DESCRIPTION:
The KetHead study is designed as a multi-center, placebo-controlled, superiority randomized controlled trial with two parallel groups and blinding of participants and outcome assessors. It will be conducted at two chronic pain centers, Toronto Western Hospital and Sinai Health System. Eligible patients will be identified and enrolled in the pain clinics. Randomization will take place upon patient enrollment. Treating physicians, patients, close contacts, study coordinators and primary outcome assessors will be blinded to treatment allocation.

Interventions common to both arms Participating patients will receive the infusion at the pain infusion unit at Toronto Western Hospital, under hemodynamic monitoring, supervised by an Anesthesiologist. At the start of the infusion, all patients will receive IV midazolam 0.04 mg.kg-1 (maximum 3 mg) and subsequently 0.01-0.02 mg.kg-1 every hour to keep participants in a sedated but arousable state (Ramsay Sedation Scale score 3 or 4)22 to blind the participants and assessors to group allocation. Eight mg of ondansetron and 8 mg of dexamethasone will be administered to all participants to prevent nausea, 5000 units of heparin will be given subcutaneously to prevent thrombo-embolic events. Medications will be administered by an Anesthesiologist.

A. Intervention group: For individuals randomized to the IV Ketamine group, 1 mg.kg-1 bolus will be given. This will be prepared as a syringe of 10 cc of Ketamine 10 mg/ml. This is followed by an infusion of 1 mg.kg-1.hour-1 (ketamine diluted in saline to 2 mg/mL at 0.5 mL.kg-1.hour-1) for six hours.

B. Control group: For individuals in the saline infusion group, an IV bolus of 0.9% saline will be given. The volume will be the same as that of the ketamine bolus for that weight, to prevent unblinding of participants and assessors. This will be followed by an infusion 0.5 mL.kg-1.hour-1 of saline for six hours. The rate of the infusion will be the same as that of a ketamine infusion for that weight to prevent unblinding of participants and assessors.

Study personnel will assess patient and collect data throughout their enrollment in the study.

During the trial, patients will be instructed to use a pain and migraine diary for collection of migraine days, pain scores and rescue pain medication during the 12 weeks after infusion.

Patients will be assessed for collection of outcomes immediately after the infusion and at 1-month, 2-months and 3-months after infusion.

Participants in both arms will wear the actigraphy device starting on the day of infusion for one month to longitudinally assess the impact of the study treatments on sleep and activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. CDH diagnosis preceding trial enrollment with headache episodes lasting for 4 or more hours occurring on 15 or more days in a month for 3 or more months (International Headache Society-IHS criteria)
3. Normal liver and kidney function tests

Exclusion criteria:

1. Pregnant or breastfeeding patients
2. Pre-existing renal impairment
3. Pre-existing liver impairment
4. Chronic benzodiazepine or antipsychotic medication use
5. History of cerebrovascular event
6. Significant and untreated hypertension or severe cardiac condition
7. Hypothyroidism
8. Glaucoma
9. Concomitant use of strong CYP2B6 or CYP2C8 inhibitor
10. Allergy or intolerance to ketamine
11. Pheochromocytoma
12. Any significant cognitive or language barriers that impede participation
13. CGRP antagonist use in 1 month or Onabotulinum-toxin A 3 months before infusion
14. Active diagnosis of Post-Traumatic Stress Disorder (PTSD)
15. Active diagnosis of Substance Use Disorder
16. Patients taking opioid medications with daily Oral Morphine Equivalents ≥80 mg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in headache days between the 2 groups | At 4 weeks
  Between-group difference in the number of headache days in the first 4 weeks after the infusion.
  (Defined as a day in which the headache lasts 4 or more hours, or a headache of any duration for which abortive treatment (anti-inflammatories, triptans, ergot derivatives, opioids) are taken. Patients will be asked to keep track of their headache days in a diary)

SECONDARY OUTCOMES:
Impact of ketamine on headache intensity after infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on headache intensity at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using Numerical Rating Scale (0-10)
Impact of ketamine on headache frequency after infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on headache frequency at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, as number of headache episodes per day
Impact of ketamine on headache duration after infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on duration of headache at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, from the headache diary maintained by patient
Impact on sleep efficiency after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on efficiency of sleep at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, measured with an actigraphy device
Impact on quality of sleep after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on quality of sleepat one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, assessed with the PSQI (Pittsburgh Sleep Quality Index) questionnaire
Impact on physical activity after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on physical activity at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, measured with actigraphy device
Impact after ketamine infusion on daily activity | At 1 month, 2 months and 3 months
  Impact of ketamine on seven daily activities (e.g. general activity, walking, mood etc.) at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, measured with Brief Pain Inventory (BPI) scale
Impact of on emotional well being (for catastrophizing) after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on emotional well being at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using the PCS (pain catastrophizing scale) scale
Impact of on emotional well being for anxiety after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on emotional well being at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using anxiety (GAD7- Generalized Anxiety Disorder-7) scale
Impact of on emotional well being for depression after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on emotional well being at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using depression (PHQ9-Patient Health Questionnaire9) questionnaire
Impact of ketamine infusion on patient satisfaction | At 1 month, 2 months and 3 months
  Impact of ketamine on patient satisfaction at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using global improvement (PGIC) scales
Impact on quality of life after ketamine infusion | At 1 month, 2 months and 3 months
  Impact of ketamine on quality of life at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using EQ-5D (European Quality of life) questionnaire
Impact of ketamine infusion on analgesic consumption | At 1 month, 2 months and 3 months
  Impact of ketamine on analgesic consumption at one month (4 weeks), two month (week 5-8) and three month (week 9-12) month after infusion, using name and dose of the analgesic use
Side effects after ketamine infusion | Immediately after infusion and after 1 week
  Side effects after the ketamine infusion as assessed using Bowdle questionnaire
Side effects after ketamine infusion | Immediately after the infusion
  Dissociative side effects assessed after the ketamine infusion, using the CADSS (Clinician Administered Dissociative States Scale) checklist

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Study results will first be disseminated at the local, national and international conferences and submitted for publication in a peer-reviewed journal.

REFERENCES:
- [Result] Schwenk ES, Dayan AC, Rangavajjula A, Torjman MC, Hernandez MG, Lauritsen CG, Silberstein SD, Young W, Viscusi ER. Ketamine for Refractory Headache: A Retrospective Analysis. Reg Anesth Pain Med. 2018 Nov;43(8):875-879. doi: 10.1097/AAP.0000000000000827. PMID 29923953
- [Result] Pomeroy JL, Marmura MJ, Nahas SJ, Viscusi ER. Ketamine Infusions for Treatment Refractory Headache. Headache. 2017 Feb;57(2):276-282. doi: 10.1111/head.13013. Epub 2016 Dec 27. PMID 28025837
- [Result] Orhurhu V, Orhurhu MS, Bhatia A, Cohen SP. Ketamine Infusions for Chronic Pain: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesth Analg. 2019 Jul;129(1):241-254. doi: 10.1213/ANE.0000000000004185. PMID 31082965
- [Derived] Hoydonckx Y, Singh M, Gilron I, Khan J, Narouze S, Dahan A, Curtis K, Cao X, Kara J, Bhatia A. Trial protocol for a multicenter randomized controlled trial to assess the efficacy and safety of intravenous ketamine for chronic daily headaches: the "KetHead" trial. Trials. 2023 Mar 1;24(1):155. doi: 10.1186/s13063-023-07186-3. PMID 36855160